CLINICAL TRIAL: NCT01954485
Title: Histological Differences in the Adhesion of Connective Tissue Around Laser-treated Abutments and Standard Abutments for Dental Implants - Clinical Trial in Humans
Brief Title: Adhesion of Connective Tissue Around Laser-treated Abutments for Dental Implants - Clinical Trial in Humans
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Barcelona (Other)
Collaborators: BioHorizons, Inc. (Industry)
Responsible Party: Principal Investigator, Raul Ayuso Montero, D.D.S., Physical Doctor, Doctor in Dental Science, University of Barcelona
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Basic Science
Other Study IDs: Laser-Lok® abutment
Record Dates: First submitted 2013-09-19; First posted 2013-10-01 (Estimated); Last update posted 2013-10-01 (Estimated); Status verified 2013-09

CONDITIONS: Periimplantitis
Keywords: LaserLok, connective tissue, adhesion
MeSH Terms: conditions — Peri-Implantitis; Tissue Adhesions

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- LaserLok abutment (Experimental): Laser microtexturing dental implant abutment
  Interventions: Procedure: Dental implant placement with a final prosthetic abutment
- 3inOne abutment (Active Comparator): Standard dental implant abutment
  Interventions: Procedure: Dental implant placement with a final prosthetic abutment

INTERVENTIONS:
Procedure: Dental implant placement with a final prosthetic abutment

SUMMARY:
This study aims to demonstrate the histological differences in the connective tissue surrounding laser-treated abutments and untreated abutments in humans.

Working hypothesis: There are differences in the adhesion of collagen fibres around implant abutments with laser-produced microgrooves and standard abutments.

DETAILED DESCRIPTION:
All patients will receive both abutment systems. The assignment of the abutments to each of the implants will be made randomly using SPSS 15.0 (SPSS Inc., Chicago, Il, United States) software.

ELIGIBILITY:
Inclusion Criteria:

* patient must have partial edentulism of at least 2 teeth
* patients that have scheduled treatment for the placement of at least 2 implants
* patients with favourable attached gingiva
* patients without systemic diseases that would prevent the emplacement of implants
* patient must accept participation in the study by signing an informed consent form

Exclusion Criteria:

* smokers of 1 or more cigarettes per day
* patients who suffer from any known condition that could be an absolute or relative contraindication to dental implant placement
* patients requiring any additional surgical technique for bone or gum graft in order to insert the dental implant
* patients who refuse to be included in the study or do not sign the informed consent form

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Dates: Start 2013-01; Primary Completion 2013-09 (Actual); Study Completion 2014-09 (Estimated)

PRIMARY OUTCOMES:
Connective tissue adhesion | 3 months
  At 90 days after the first operation, a second surgical procedure will be scheduled. A cilindrical scalpel of a diameter 2 mm greater than the abutment is used to make the incision and the abutment unscrewed together with the gingival insertion surrounding it for histological study.
  The attachment of connective tissue to the abutments will be determined by microscopic observation. It will be a binary variable: attachment IS present (YES-A); attachment IS NOT present (NO-A).

CONTACTS AND LOCATIONS:
Overall Officials: Monica Blazquez-Hinarejos, DDS, Principal Investigator — Barcelona University; Raul Ayuso-Montero, DDS, PhD, Study Director — Barcelona University; Jose Lopez-Lopez, MD, PhD, Study Chair — Barcelona University; Cristina Manzanares-Cespedes, MD, PhD, Study Director — Barcelona University
Locations (1):
- Hospital Odontològic, L'Hospitalet de Llobregat, Barcelona, Spain